CLINICAL TRIAL: NCT06206356
Title: Lumbar Injectrode Feasibility Evaluation
Acronym: LIFE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuronoff, Inc (Industry)
Collaborators: Ohio Pain Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NCP-11
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Chronic Pain; Lower Back Pain Chronic
Keywords: Neuromodulation; Injectable Electrode; Medical Device Safety; Injectrode; Healthy Volunteer
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- PNS Injectrode F1 (Experimental)
  Interventions: Device: PNS Injectrode F1

INTERVENTIONS:
Device: PNS Injectrode F1 — The PNS Injectrode F1 is a flexible conductor that conforms to the shape of a peripheral nerve and patient anatomy. The device is approximately 1 mm in overall diameter and is provided in lengths of 9 or 10 cm. The device is placed in a minimally invasive procedure via a standard 18g needle. The stimulating end of the device is placed in close proximity to the lumbar medial branch nerve with a collector end left subcutaneously. Electrical stimulation is provided via an externally placed patch electrode connected to the provided external pulse generator over the collector end of the device. Transcutaneous electrical stimulation will occur prior to device placement, on Day 0 after device placement, and on Day 25 prior to device removal. Minimally invasive removal is completed by a small incision and forceps using standard medical procedures and equipment.
  Other Names: Injectrode

SUMMARY:
The goal of this non-significant risk study is to determine whether stimulation with transcutaneous waveforms applied on the outside of the body and subcutaneously conducted to the lumbar medial branch nerve elicits visible (via ultrasonic imaging) or palpable multifidus muscle activation within the short-term (<28 day) placement of the Neuronoff PNS Injectrode F1 in healthy volunteers.

The main questions it aims to answer are:

* Can the PNS Injectrode F1 be safely inserted on the lumbar medial branch nerve for up to 28 days?
* Can the PNS Injectrode F1 be safely used to stimulate the lumbar medial branch nerve to activate the multifidus muscle?

Participants will

* Receive transcutaneous stimulation of the lower back prior to device placement, after device placement, and prior to explant
* Insert the PNS Injectrode F1 device on the lumbar medial branch nerve
* Have the device inserted for up to 28 days and then explanted
* Visit Schedule: Screening/Enrollment, Day 0, Day 2 (email), Day 25, 2 Days Post Explant (email), Day 35

ELIGIBILITY:
Inclusion Criteria:

* Be 21 years of age or older when written informed consent is obtained.
* Literate, able to speak English and able to complete questionnaires independently.
* Willing to sign an Institutional Review Board (IRB)-approved informed consent form (ICF) and deemed capable of complying with the study requirements.
* Are currently receiving optimal medical management and considered medically stable as judged by the investigator for any significant medical condition.
* Be able to tolerate minimally invasive electrical stimulation.
* Be willing and able to understand and comply with all study-related procedures during the course of the study, and attend all scheduled study visits.

Exclusion Criteria:

* Severe cognitive impairment as determined by the Investigator.
* If female and sexually active, and the subject is not using a reliable form of birth control, is not surgically sterile or at least two years post-menopausal, the subject shall be excluded, as confirmed by the Investigator.
* If female, have a positive pregnancy test at the screening and/or Day 0 visit.
* Pre-existing motor, balance, proprioception, or sensory deficits as determined by Investigator.
* Show symptoms indicative of Covid-19 as assessed during enrollment.
* Have a skin condition at the planned surgical location.
* Have a blood coagulation disorder or other indication with the potential to impact the study biocompatibility data in unpredictable ways.
* Have a medical condition that is a contraindication for minimally invasive procedures.
* Have a cardiac demand pacemaker, implanted defibrillator or another implanted electronic device.
* Have a history of cardiac arrhythmia with hemodynamic instability.
* Be implanted with a neurostimulator.
* Have any active electrical implant of any other kind.
* Have an active infection.
* Current coagulopathy, thrombocytopenia or bleeding diathesis (confirmed by clinical history and, if clinically indicated, by coagulation screening).
* Have untreated drug habituation or dependence.
* Have uncontrolled seizures (averaging > 2 seizures per month).
* Currently require, or be likely to require, diathermy and/or MRI during study duration.
* Known hypersensitivity to any of the procedural agents or materials in the study device that is inserted into the subject.
* Have a history of adverse reactions to local anesthetics (e.g. lidocaine).
* A systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study (e.g. current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction, uncontrolled diabetes, etc.).
* Any experimental drug or device used within 30 days prior to the screening visit or during the course of the clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Device Effects (SADEs) | 35 days
  The safety endpoint will be the percentage of subjects that experience serious adverse device effects (SADE).
Proportion of Subjects with Multifidus Muscle Activation as determined by PI via Ultrasound Imaging and Palpation | 25 days
  The efficacy endpoint will be the proportion of subjects with a clinically meaningful activation of the multifidus muscle(s) unilaterally or bilaterally utilizing transcutaneous stimulation on Day 0 and on or before the Day 25 visit. Meaningful activation will be evaluated by the PI based on ultrasonic imaging as well as palpation.

CONTACTS AND LOCATIONS:
Overall Officials: Amol Soin, MD, MBA, Principal Investigator — The Ohio Pain Clinic
Locations (1):
- The Ohio Pain Clinic, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No